CLINICAL TRIAL: NCT03533621
Title: The Effect of Probiotics on Gut Microbiome and Adiposity
Brief Title: Gut Microbiome, Adiposity, and Probiotics (GMAP)
Acronym: GMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Rady Children's Hospital (Unknown)
Responsible Party: Principal Investigator, Kay Rhee, Associate Professor of Pediatrics, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 141045
Record Dates: First submitted 2018-04-18; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Subjects were randomized to probiotic or placebo group, and remained in that group for the 12 week study period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-control trial. Investigators, subjects, and assessors were unaware of which group they were randomized to. Subjects received pills in a paper bad that looked identical to each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): 1 Probiotic pill, twice a day, for 12 weeks + 20 min weekly support to increase fruit and vegetable consumption
  Interventions: Dietary Supplement: Probiotic - VSL#3
- Placebo (Placebo Comparator): 1 placebo pill (soy protein powder), twice a day, for 12 weeks + 20 min weekly support to increase fruit and vegetable consumption
  Interventions: Dietary Supplement: Placebo pill - soy protein powder

INTERVENTIONS:
Dietary Supplement: Probiotic - VSL#3 — Subjects received a weekly supply of pills for 12 weeks along with support to change their diet to consume more fruits and vegetables. Subjects met with an interventionist weekly to report on pill consumption, stool changes, and get help with changing their dietary behaviors
  Arms: Probiotic
Dietary Supplement: Placebo pill - soy protein powder — Subjects received a weekly supply of pills for 12 weeks along with support to change their diet to consume more fruits and vegetables. Subjects met with an interventionist weekly to report on pill consumption, stool changes, and get help with changing their dietary behaviors
  Arms: Placebo

SUMMARY:
Recent studies have shown that the bacteria in the gut (gut microbiome) can affect adiposity levels and inflammation. In animal studies, changing these bacteria has been linked with decreased fat mass and inflammation as well as improved metabolism. Probiotics can be a safe method of altering the gut microbiome in humans and have shown promising results in adults with regards to changing adiposity and inflammatory markers. However, it may also be important to provide the right dietary milieu (i.e. high fruit and vegetable/low saturated fat diet) in order to see the benefits of probiotics on these physiologic markers. At this time, no one has offered probiotics in the context of the right dietary milieu and tested it in children. This pilot proposal is innovative because it will be the first to test how well probiotics work in the context of a diet high in fruits and vegetables to change the gut microbiome, decrease fat mass, and improve inflammatory markers in overweight/obese children. This protocol will allow one to better understand the effect of probiotics on these physiologic functions and determine acceptability and feasibility of taking daily probiotics.

DETAILED DESCRIPTION:
The goal is to study the effect of probiotics on changing the gut microbiome of overweight/obese children. Since there appears to be a diet-by-microbiota interaction for optimal effects on adiposity, it will be important to administer the probiotics within the context of increased fruit/vegetable (F/V) intake and decreased fat intake. Because changes in diet alone can also induce changes in the gut microbiota, this study will use a double-blind, randomized, placebo-control design to determine whether changes in gut microbiota are greater with the addition of probiotics (High F/V diet + Probiotics) compared to diet alone (High F/V diet + Placebo). The primary aim is to test the effect of these 2 arms on changing the gut microbiota, fat mass, and inflammation in children. The study will also examine the acceptability of taking probiotics and changes in other physiologic measures.

The Specific aims of this proposal are:

1. To examine the effect of diet high in F/V +/- probiotics on change in gut microbiota, adiposity, and inflammation (measured by C-reactive protein, TNF-a, and IL-6);
2. To examine the effect of diet high in F/V +/- probiotics on physiologic measures including blood pressure, fasting insulin and glucose, and adiponectin;
3. To determine the acceptability and feasibility of taking daily probiotics over a 12 week period.

ELIGIBILITY:
Inclusion Criteria:

* BMI >= 85th percentile
* 7-16 years old
* parent willing to participate

Exclusion Criteria:

* 1) taking any oral or topical antibiotics or probiotics within the last month prior to the start of the intervention, 2) allergy to milk or milk products, 3) taking any diabetes medication, lipid-lowering drugs, or anti-inflammatory drugs, 4) be immune compromised; 5) 5% weight change or greater within the last three months, 6) psychiatric or medical illness that would hinder their ability to participate in weekly sessions, 7) receiving treatment for a major psychiatric disorder, including an eating disorder, 8) developmental delay such that the intervention materials will not be appropriate, and 9) the possibility of moving out of the area within the time frame of the study.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Adiposity | 12 weeks
  change in total % fat mass as measured by DXA scan measured at baseline (week 0) and study completion (week 12)
hsCRP | 12 weeks
  high sensitivity C-reactive protein (mg/L) measured at baseline (week 0) and study completion (week 12)
IL-6 | 12 weeks
  Interleukin 6 (pg/ml) measured at baseline (week 0) and study completion (week 12)
TNF-alpha | 12 weeks
  Tumor necrosis factor alpha (pg/ml) measured at baseline (week 0) and study completion (week 12)
Adiponectin | 12 weeks
  adiponectin (ug/ml) measured at baseline (week 0) and study completion (week 12)
Acceptability of taking pills | week 12
  Acceptability of taking pills daily for 12 weeks assessed with 3 separate questions: Did your child take his/her pill daily (1 = not at all, 3 = sometimes, 5 = every day); Did your child have trouble remembering to take his/her pill daily (1 = not at all, easy to remember, 5 = had a lot of trouble remembering); Did your child like taking his/her pill (1 = not at all, 5 = loved it!). Parents were asked to complete these questions at study completion (week 12). The second question will be reverse-scored, and higher scores will indicate better acceptability. Each question will be viewed as separate items, and not combined to create a summary score.
Proportion of participants with side effects | 12 weeks
  weekly assessment of any side effects reported by participants including nausea, abdominal pain, bloating, or skin reactions

SECONDARY OUTCOMES:
Bristol Stool chart | 12 weeks
  changes in stooling pattern as assessed by the Bristol Stool Chart, measured at baseline (week 0), weekly during the study (weeks 1-11), and study completion (week 12)
gut microbiome | 12 weeks
  Changes in the composition and alpha and beta diversity of the gut microbiome using 16SrRNA amplicon sequencing. DNA sequencing will be performed using MiSeq platforms. Samples were obtained at baseline (week 0) and study completion (week 12).

IPD SHARING:
Plan to Share IPD: No